CLINICAL TRIAL: NCT05659966
Title: NEW Soul D&I: Expanding the Reach of the Nutritious Eating With Soul (NEW Soul) Program
Brief Title: Nutritious Eating With Soul Dissemination and Implementation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00116789
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Nutrition, Healthy; Eating Behavior
MeSH Terms: conditions — Feeding Behavior | interventions — Diet, Plant-Based

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention condition participants will be instructed to follow a plant-based diet. The intervention participants will receive weekly group classes for 3 months at a local restaurant and will receive guidance on how to choose foods to meet their nutrient needs that fit within the vegan diet. The intervention participants will receive a voucher each week for a free plant-based meal at the restaurant.
  Interventions: Behavioral: Plant-based diet
- Control (Active Comparator): Participants in the active control condition will receive meal vouchers to the restaurant. The active control condition participants will not receive any instruction to follow a particular diet or support. Participants in this condition will receive all intervention material and attend a class at the end of the study to learn about the intervention diet.
  Interventions: Other: Voucher only

INTERVENTIONS:
Behavioral: Plant-based diet — Participants will receive a behavioral intervention on a plant-based diet in partnership with a local restaurant.
  Arms: Intervention
Other: Voucher only — Participants will receive vouchers to a local restaurant. Participants will not attend nutrition classes but will receive a class at the end of the 12-week study.
  Arms: Control

SUMMARY:
The investigators will conduct a full dissemination and implementation study using a type 2 hybrid effectiveness-implementation design. The investigators will conduct this study in the community and work with two vegan soul food restaurants. The investigators propose to examine the effectiveness and implementation of community-delivered, 3-month NEW Soul program among participants (N=228).

Using a randomized design, the investigators will assess effectiveness of two delivery approaches: (1) In-person, live weekly classes with restaurant vouchers (intervention) or (2) restaurant voucher-only (active control).

The investigators will also conduct a cost-effectiveness analysis of delivering the online intervention plus voucher vs. voucher-only with the outcome of cost/change in weight, healthy eating index, and quality adjusted life year.

Lastly, the investigators will examine the implementation of the NEW Soul study with participants and intervention staff.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as African American
* Be between the ages of 18-65 years
* Body Mass Index between 25- 49.9 kg/m2
* Able to travel to restaurant for classes
* Be able to attend all monitoring and weekly class visits
* Be willing to be randomized to either group

Exclusion Criteria:

* Currently following a plant-based diet
* Diagnosed with diabetes that is controlled by medication
* Currently pregnant or breastfeeding (or plan to become pregnant in the next 24 months)
* Under the age of 18 years old
* Over the age of 65 years old
* Currently participating in a weight loss program
* Has lost more than 10 pounds in the past 6 months
* Potential eating disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in body weight | 3-months
  Changes in body weight in kilograms
Changes in diet quality | 3-months
  Changes in dietary quality as assessed by the Healthy Eating Index

SECONDARY OUTCOMES:
Cost-effectiveness | 3-months
  The investigators will assess the costs between delivering the in-person intervention plus voucher vs. voucher-only with the outcome of cost per change in participant body weight, healthy eating index score, and quality adjusted life year (QALY). The cost-effectiveness evaluation will also include estimating costs of the intervention itself (e.g., training, delivery, infrastructure).
Implementation | 3-months
  Implementation will be assessed using qualitative data collection with participants via focus groups and restaurant staff leading the intervention via in-depth interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- Mimsy's Restaurant, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, data will be shared with other researchers. Data will not be publicly available to protect participant confidentiality. The informed consent document will include information that de-identified data may potentially be shared with other researchers.
Supporting Information: Study Protocol
Time Frame: Upon reasonable request, participant data will be shared with other researchers.
Access Criteria: If granted, a password protected file with de-identified data of participants will be shared with other researchers.